CLINICAL TRIAL: NCT02219009
Title: A Multicenter, 8-week, Open-label Study to Assess Usability of the Medical Information Device #1 (MIND1) System in Adult Subjects With Schizophrenia Who Are Treated With Oral Aripiprazole
Brief Title: Open-label Study to Assess Usability of the Medical Information Device #1 (MIND1) System in Adults With Schizophrenia On Oral Aripiprazole
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 316-14-220
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Schizophrenia; Mental Disorder; Nervous System Diseases
Keywords: OPC-14597 Digital; Aripiprazole; Medical Information Device #1 System (MIND1); Treatment Adherence; Ingestible Event Marker
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Nervous System Diseases; Treatment Adherence and Compliance

ARMS (1):
- MIND1 System (Experimental)
  Interventions: Device: MIND1 System

INTERVENTIONS:
Device: MIND1 System — Subjects will receive aripiprazole tablets embedded with an IEM. They will discontinue their normally prescribed oral aripiprazole tablets and will take the aripiprazole + IEM tablets (eg, at the previously prescribed dose) during the 8-week treatment period for this study. Aripiprazole + IEM tablets must be taken on a once-daily dosing schedule.
  Other Names: OPC-14597 Digital

SUMMARY:
The purpose of this study is to determine the usability of the Medical Information Device #1 (MIND1) system in adults with schizophrenia who are treated with oral aripiprazole.

DETAILED DESCRIPTION:
Poor adherence to medication is a well-recognized problem in psychiatric patients. Although a variety of treatment models have been developed to improve management of patients in general and medication adherence in particular, poor medication adherence remains a major barrier to achieving optimal health.

The MIND1 System includes a drug-device combination, a patch, and application software to convey level of activity and rest and to mark events through the act of ingestion.

The purpose of this open-label study is to determine the usability of the Medical Information Device #1 (MIND1) System in adults with schizophrenia. Approximately 32 subjects with schizophrenia, between 18 and 65 years of age (inclusive) who are currently prescribed and stabilized on oral aripiprazole, will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be prepared and able to give written (signed and dated) informed consent, which includes adherence to study requirements and restrictions before enrolling in the study. Subjects must be willing to adhere to study procedures, including troubleshooting of the MIND1 System by a third party if needed (third party will be blinded to personal health information).
* Male and female subjects 18 to 65 years of age, inclusive, at time of informed consent.
* Subjects who have a primary current diagnosis of schizophrenia, as defined by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria. Subjects may be symptomatic at screening, but must be able to be treated as outpatients.
* Subject is cooperative, able to ingest oral medication, and willing to complete all aspects of study.
* Subject is currently prescribed oral aripiprazole for schizophrenia at one of the following single daily doses (10, 15, 20, or 30 mg), and is deemed likely to remain on this same stable dose throughout the course of the study. Subject has not had any changes in their aripiprazole regimen or dose over the 2 weeks before screening.
* Subject must be able and willing to carry the MIND1 System smartphone on his/her person and complete all tasks, as well as adequately operate all devices, as applicable. Caregiver or other third-party assistance can be utilized, if needed, although all subjects should be encouraged to attempt all tasks themselves.
* Subject likely possesses the capacity to utilize the technology interfaces (eg, open and navigate software applications using the touch screen) and telephone features of a smartphone. The subject has satisfactory mobile phone reception (preferably 3 bars or more, or have Wi-Fi) at home and/or at work for study-designated wireless carrier.
* Subject is not pregnant or breast-feeding, and does not plan to become pregnant.
* Skin on the anterior chest just above the lower edge of the rib cage that is free of any dermatological problems (eg, dermatosis or dermatitis, open wounds, or other skin disorders such as warts, rashes, atopic dermatitis, or irritations).

Exclusion Criteria:

* Subjects with a current DSM-5 diagnosis other than schizophrenia, including major depressive disorder, bipolar disorder, schizoaffective disorder, delirium, major neurocognitive disorder (eg, dementia), intellectual developmental disorder, or any other diagnosis that might impact the subject's ability to participate in the study. Other disorders that are not the focus of treatment and will not impact the subject's ability to participate in all aspects of the study (eg, social anxiety disorder) may be included.
* Subjects with a current DSM-5 diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder.
* Subjects who exhibit prominent negative symptoms that, in the judgment of the investigator, will interfere with study procedures or unable to adhere with study requirements.
* Subjects who are currently on a long-acting injectable antipsychotic.
* Subjects who are likely to be incapable of using the MIND1 System technology, even with assistance.
* On the Columbia-Suicide Severity Rating Scale (C-SSRS) Subjects who answer "Yes" to Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) and whose most recent episode meeting criteria for this C-SSRS Item 4 occurred within the last 3 months, OR Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) and whose most recent episode meeting criteria for this C-SSRS Item 5 occurred within the last 3 months, OR Subjects who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred within the last 1 year, OR Subjects who, in the opinion of the investigator, present a serious risk of suicide.
* Subject has received any investigational product within the last 30 days, including the MIND1 System (eg, subjects who participated in Cohort 1 of this study are not eligible for Cohort 2).
* Subjects who have a history or evidence of a medical condition that would expose them to an undue risk of a significant AE or interfere with assessments of safety or usability during the course of the study, including but not limited to, hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, hematologic, or immunologic disease, as determined by the clinical judgment of the investigator.
* Subjects with epilepsy or a history of seizures (except for a single childhood febrile seizure, post traumatic seizure, alcohol withdrawal seizure, etc).
* Subjects with a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia, as assessed by the investigator.
* Subjects who are known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones.
* Subjects with a history of hypersensitivity to antipsychotic agents.
* Subjects with a known allergy to adhesive tape or any pertinent components of the patch or IEM
* Sexually active women of childbearing potential who will not commit to utilizing 2 of the approved birth control methods or who will not remain abstinent during this study and for 30 days following the last dose of study medication.
* Sexually active males (unless sterile, defined as having had a bilateral orchiectomy) who will not commit to utilizing 2 of the approved birth control methods or who will not remain abstinent during the study and for 90 days following the last dose of study drug.
* Subject has a current history (within the past month) of a substance use disorder (excluding tobacco) which meets DSM-5 criteria, or demonstrates a positive result on the urine drug test during screening. Subjects with a positive drug screen for drugs of abuse (excluding cannabinoids) are excluded and may not be retested or rescreened. Subjects with a positive urine drug screen resulting from use of prescription (such as opioids) or over-the-counter medications or products that, in the investigator's documented opinion, do not signal a clinical condition that would impact the safety of the subject or interpretation of the study results may continue evaluation for the study following consultation and approval by the Medical Monitor.
* Subjects who, in the opinion of the investigator, are acutely psychotic or who exhibit symptoms currently requiring hospitalization.
* Subjects unwilling to refrain from the use of topical products on the skin patch sites.
* Subjects unwilling or unable to complete the evaluations included in this study, which include audio recording of the subject's voice and require the ability to distinguish colors (eg, subjects unwilling to be recorded and colorblind subjects are to be excluded from participation in this study)
* Any subject who, in the opinion of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Peters-Strickland, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (6):
- United States (6):
  - Cerritos, California
  - Garden Grove, California
  - Oceanside, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - St Louis, Missouri

REFERENCES:
- [Derived] Jan M, Coppin-Renz A, West R, Gallo CL, Cochran JM, Heumen EV, Fahmy M, Reuteman-Fowler JC. Safety Evaluation in Iterative Development of Wearable Patches for Aripiprazole Tablets With Sensor: Pooled Analysis of Clinical Trials. JMIR Form Res. 2023 Dec 12;7:e44768. doi: 10.2196/44768. PMID 38085556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 67 participants at 6 trial sites in the United States.
Pre-assignment Details: The trial included a screening period (≤ 2 weeks), a treatment period (8 weeks), and a safety follow-up period (2 weeks). Participants enrolled under the original version of the protocol were considered to comprise a first cohort (Cohort 1), while subjects enrolled under Amendment 1 were considered to comprise a separate second cohort (Cohort 2).
Groups:
- MIND1 System (Cohort 1): Participants received aripiprazole tablets embedded with an ingestible event marker (IEM). They discontinued their normally prescribed oral aripiprazole tablets and took aripiprazole + IEM tablets (eg, at the previously prescribed dose) during an 8-week treatment period. Aripiprazole + IEM tablets were taken on a once-daily dosing schedule. Participants wore a patch which received signals from the IEM and transmitted information to a Medical Data Device System (MDDS).
  Cohort 1 participants were enrolled under the original protocol.
- MIND 1 System (Cohort 2): Participants received aripiprazole tablets embedded with an IEM. They discontinued their normally prescribed oral aripiprazole tablets and took aripiprazole + IEM tablets (eg, at the previously prescribed dose) during an 8-week treatment period. Aripiprazole + IEM tablets were taken on a once-daily dosing schedule. Participants wore a patch which received signals from the IEM and transmitted information to a MDDS.
  Cohort 2 participants were enrolled under protocol amendment 1.
Period: Overall Study
Arm/Group | MIND1 System (Cohort 1) | MIND 1 System (Cohort 2)
Started | 37 | 30
Completed | 27 | 22
Not Completed | 10 | 8
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Adverse Event | 2 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol deviation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled sample - all participants who signed an informed consent and entered the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | MIND1 System (Cohort 1) | MIND 1 System (Cohort 2) | Total
Number analyzed (Participants) | 37 | 30 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (10.3) | 47.6 (8.9) | 46.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 27 | 23 | 50

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Are Able to Pair & Apply a Patch Independently & Successfully by the End of the Week 8 Study Visit as Defined by a Score of 91 to 100 on the Subject Ability to Use System Scale - Healthcare Professional Version (SAUSS-HCP)
Description: Proportion of participants who are able to pair and apply a patch independently and successfully by the end of the Week 8 study visit (or early termination, if applicable), as defined as a score of 91 to 100 on the participant's Ability to Use System Scale - Healthcare Professional Version (SAUSS-HCP). A participant was considered to have successfully and independently applied a patch if the SAUSS-HCP was at least 91 for at least one postbaseline score.
Time Frame: Baseline to Week 8
Population: The intent-to-treat (ITT) population - all participants who entered the trial and used the MIND1 system
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MIND1 System (Cohort 1) | MIND 1 System (Cohort 2)
Number analyzed (Participants) | 37 | 30
percentage of participants | 54.1 [36.9 to 70.5] | 56.7 [37.4 to 74.5]

2. Secondary Outcome: Proportion of Participants Able to Pair & Apply a Patch Successfully, Independently, or With Minimum Assistance, by the End of the Week 8 Study Visit, as Defined by a SAUSS-HCP Score of 71 to 100.
Description: Proportion of participants who are able to pair and apply a patch successfully, independently, or with minimum assistance, by the end of the Week 8 study visit (or early termination, if applicable), as defined by a Participant's Ability to Use System Scale - Healthcare Professional Version (SAUSS-HCP) score of 71 to 100. Participants were considered to have paired and applied a patch independently or with minimal assistance if their SAUSS-HCP score was at least 71 for at least one postbaseline score.
Time Frame: Baseline to Week 8
Population: ITT population - all participants who entered the trial and used the MIND1 system.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MIND1 System (Cohort 1) | MIND 1 System (Cohort 2)
Number analyzed (Participants) | 37 | 30
percentage of participants | 83.8 [68.0 to 93.8] | 80.0 [61.4 to 92.3]

3. Secondary Outcome: Proportion of Time During the Study Period When Participants Wear Their Patches
Description: Proportion of time during the study period when participants wear their patches; the time duration of patch wearing will be calculated based on digital health data. Percentage of participants' patch wearing time was calculated as (total duration a patch was worn / trial duration) x 100.
Time Frame: Baseline to Week 8
Population: ITT population - all participants who entered the trial and used the MIND1 system.
Measure: Mean (Standard Deviation); unit: % of time participants wore patch
Arm/Group | MIND1 System (Cohort 1) | MIND 1 System (Cohort 2)
Number analyzed (Participants) | 37 | 30
% of time participants wore patch | 74.4 (22.0) | 66.2 (27.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing the informed consent, throughout the 8 week treatment period and for 2 weeks after the last treatment.
Arm/Group | MIND1 System (Cohort 1) | MIND 1 System (Cohort 2)
Serious Adverse Events (participants affected / at risk) | 2/37 | 0/30
Other Adverse Events (participants affected / at risk) | 17/37 | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MIND1 System (Cohort 1) (N=37) | MIND 1 System (Cohort 2) (N=30)
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MIND1 System (Cohort 1) (N=37) | MIND 1 System (Cohort 2) (N=30)
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Increased appetitie (Metabolism and nutrition disorders) | 0 | 2
Somnolence (Nervous system disorders) | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Center may publish study results but ≥ 60 days prior to any public presentation, a copy is sent to Sponsor for review and Center can delay publication for 60 days to permit Sponsor to protect its intellectual property rights or confidential information contained within the publication. The first publication is a joint publication, if Center is part of a multi-center study. Center is free to publish, if there is no multi-center publication within 18 months of completion/ termination of study.